CLINICAL TRIAL: NCT06384677
Title: Comparison of Postoperative Analgesia Methods in Patients Undergoing Major Intraabdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 03.03.2023/371
Record Dates: First submitted 2024-04-18; First posted 2024-04-25 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-04

CONDITIONS: Abdominal Cancer; Abdomen Disease
Keywords: major abdominal surgery; M-TAPA; opioid consumption; postoperative analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M-Tapa + IV PCA applied group (Other): After appropriate skin disinfection, the transversus abdominis, internal oblique and external oblique muscles were determined with a high-frequency linear probe (Esaote) at the costochondral angle in the sagittal plane under ultrasound guidance at the 10th costal border. A 21-G, 80-mm peripheral block needle was placed in the cranial direction using the in-plane technique, the needle tip did not exceed the cranial edge of the 10th costal cartilage, and 20 ml of 0.25% bupivacaine was applied to the lower surface of the chondrium on both sides, right and left. .
  Interventions: Other: M-Tapa Block
- IV PCA applied group (Other): In the IV PCA group, the surgeon performed local infiltration with 40 mL of 0.25% bupivacaine around the incisions. All patients were provided postoperative analgesia with intravenous patient-controlled analgesia (IVHKA). When pain was expressed by the patient, the patient pressed a button and the IV HKA pump was programmed to deliver a 1 ml bolus dose with a 10-minute lockout interval and no background infusion allowed. Each 1 ml of IVHKA solution contains 1 mg of morphine.
  Interventions: Other: M-Tapa Block

INTERVENTIONS:
Other: M-Tapa Block — M-TAPA block was performed bilaterally with 20 mL of 0.2% bupivacaine under ultrasound guidance at the end of surgery

SUMMARY:
This study aims to examine the effects of M-TAPA applied for postoperative analgesia in patients who had major intraabdominal surgery on the postoperative pain score, the change in the postoperative total opioid requirement and the side effects.

DETAILED DESCRIPTION:
The investigators seperated the patients into two groups as M-TAPA applied group and control group.In group M-TAPA, M-TAPA block was performed bilaterally with 20 mL of 0.2% bupivacaine under ultrasound guidance at the end of surgery. No block was performed in the control group. The participants were administered morphine through patient controlled analgesia (PCA) pump with a bolus dose of 1 mg, 15 min lockout interval. The postoperative pain scores (the numeric rating scores (NRS)), total opiod consumption in the first 48 h, and opioid related side effects were recorded.

ELIGIBILITY:
Inclusion Criteria:

* patient > 17 years old
* ASA score 1-3
* undergoing major intra-abdominal surgery

Exclusion Criteria:

* ASA IV patients
* patients with known neurological or psychiatric disorders
* patients with clinically significant cardiovascular, respiratory, hepatic, renal or metabolic disease
* patients with long-term drug (opioid) or alcohol dependence
* patients with BMI>30
* patients with intellectual disability
* patients who developed massive bleeding and coagulopathy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | Postoperative 24 hours
  The postoperative opioid consumption

SECONDARY OUTCOMES:
NRS Scores | postoperative 24 hours
  Numeric Rating Scale score (rating from 1 to 10. 1:no pain to 10: worst pain ever)
the need for rescue analgesia | postoperative 24 hours
  if NRS>4: apply rescue analgesia: the total count of rescue analgesia need
side effects | postoperative 24 hours
  nausea- vomiting

CONTACTS AND LOCATIONS:
Overall Officials: GAMZE ÇABAKLI, Study Chair — Marmara Univercity
Locations (1):
- Marmara University Pendik Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoyme U, Baumueller A, Madsen PO. Antibiotics excretion in canine vaginal and urethral secretions. Invest Urol. 1978 Jul;16(1):35-8. PMID 29017